CLINICAL TRIAL: NCT06027333
Title: Self-efficacy and Well-being of Patients With Fibrotic Interstitial Lung Disease - an Observational Study
Brief Title: Self-efficacy and Well-being of Patients With Fibrotic Interstitial Lung Disease
Status: Recruiting | Type: Observational
Sponsor: Berner Reha Zentrum AG (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other); Zurich University of Applied Sciences (Other); University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: BernerRehaZentrum
Record Dates: First submitted 2023-08-31; First posted 2023-09-07 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Interstitial Lung Disease; Fibrotic Lung Disease; Self Efficacy; Self-management; Patient Education; Quality of Life
Keywords: self efficacy; self-management; patient education; well-beeing; quality of life; fibrotic lung disease; interstitial lung disease
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: inpatient rehabilitation — This is an uncontrolled observational study on patients undergoing usual care in pulmonary rehabilitation and care
  Other Names: outpatient consultations for interstitial lung disease

SUMMARY:
Patients with fibrotic insterstitial lung disease (ILD) participating in inpatient rehabilitation or in outpatient pulmonary care will be invited to participate in this observational study. Patients will fill out questionnaire regarding quality of life and symptoms at baseline and follow-up (at the end of rehabilitation or after the second outpatient ILD consultation). Additionally, clinical data obtained in clinical routine or for the IIP registry will be used for this project.

The aim is to assess changes in self-efficacy and quality of life over time and to establish a control cohort for a later feasibility study on a educational and self-management intervention (currently in planning).

ELIGIBILITY:
Inclusion criteria are:

* For Berner Reha Zentrum only: Diagnosis of a FILD as major indication for pulmonary rehabilitation
* For Inselspital only: Enrolled in Idiopathic interstitial Pneumonia (IIP) cohort study (Nr. 246/15 / PB_2016-01524) and agreed to further use of data for further research purpose
* Age ≥ 18 years
* Written informed consent

Exclusion criteria are:

* Cognitive inability or insufficient knowledge of project language (German) to follow informed consent or study procedures
* Sarcoidosis

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with fibrotic lung disease participating in an inpatient rehabilitation or in outpatient consultations for interstitial lung disease
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in Self-efficacy | From t0 to t2 (60-120 days after t0)
  Pulmonary Rehabilitation Adapted Index of Self-Efficacy (PRAISE) tool

SECONDARY OUTCOMES:
Change in Self-efficacy | From t0 to t1 (14-40 days after t0)
  Pulmonary Rehabilitation Adapted Index of Self-Efficacy (PRAISE) tool
Change in health related quality of life | From t0 to t1 (14-40 days after t0) and from t0 to t2 (60-120 days after t0)
  King's Brief Interstitial Lung Disease (K-BILD) health status questionnaire,
Change in functional status | From t0 to t1 (14-40 days after t0) and from t0 to t2 (60-120 days after t0)
  King's Brief Interstitial Lung Disease (K-BILD) health status questionnaire,
Change in self-reported health status | From t0 to t1 (14-40 days after t0) and from t0 to t2 (60-120 days after t0)
  EQ-VAS Score [0 -100] (worst to best health status)
Change in self-reported symptoms | From t0 to t1 (14-40 days after t0) and from t0 to t2 (60-120 days after t0)
  Leicester Cough Questionnaire
Change in self-reported anxiety and depression | From t0 to t1 (14-40 days after t0) and from t0 to t2 (60-120 days after t0)
  Hospital Anxiety and Depression Scale [0-21] (high number indicates high symptoms)
Symptom Visual Analog Scales | From t0 to t1 (14-40 days after t0) and from t0 to t2 (60-120 days after t0)
  Visual Analog Scales [0-100] for Cough, Dyspnoea, Fatigute, Emotions to self-report severity, impairement and self-efficacy in symptom management. (100 means high severity, high impairment and high self-efficacy)
Supplemental oxygen needs for activity and at rest | t0, t1 (14-40 days after t0) and t2 (60-120 days after t0)
  routinely collected data
Re-hospitalization and survival | from t0 to t2 (60-120 days after t0)
  routinely collected data

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Berner Reha Zentrum, Rehabilitation & Sports Medicine, Insel Group, University Hospital Berne, Bern, Heiligenschwendi
  - Department of Pulmonary Medicine, Inselspital, Bern University Hospital, University of Bern, Bern

IPD SHARING:
Plan to Share IPD: Undecided